CLINICAL TRIAL: NCT00352170
Title: Calcium and Vitamin D Malnutrition in Elderly Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Joan M. Lappe, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ag14683
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Osteoporosis; Secondary Hyperparathyroidism
Keywords: calcium; vitamin D; secondary hyperparathyroidism; osteoporotic fractures
MeSH Terms: conditions — Osteoporosis; Hyperparathyroidism, Secondary; Osteoporotic Fractures | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): calcium supplementation
  Interventions: Dietary Supplement: calcium supplementation
- 2 (Experimental): calcium and vitamin D3 supplementation
  Interventions: Dietary Supplement: calcium and vitamin D3 supplementation
- 3 (Experimental): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: calcium supplementation — calcium carbonate 1500 mg/day
  Arms: 1
Dietary Supplement: calcium and vitamin D3 supplementation — calcium carbonate 1500 mg/day vitamin D3 1000 IU/day
  Arms: 2
Dietary Supplement: Placebo — calcium and vitamin D3 placebo
  Arms: 3

SUMMARY:
This study is designed to test whether calcium supplementation alone or calcium plus vitamin D reduces the incidence of fractures, reduces high parathyroid secretory activity, and halts bone loss in a population-based sample of women 55+ years of age.

* A calcium supplement of 1400 mg/d will significantly reduce the cumulative incidence of spine and appendicular fractures over four years for independently living, rural women 55 years of age and older compared to similar women on their usual diets.
* A calcium supplement of 1400 mg/d plus 1100 IU vitamin D/d will significantly reduce the cumulative incidence of spine and appendicular fractures compared to a calcium supplement only.

DETAILED DESCRIPTION:
We are conducting a 4-year randomized, double-blind, placebo controlled trial of calcium or calcium with vitamin D supplementation. We randomly sampled the population of healthy, independent living women 55+ years in nine rural counties. We randomly assigned 1180 women to one of three groups: Group 1 receives calcium (1400 mg/d) and vitamin D placebo, Group 2 receives both calcium (1400 mg/d) and vitamin D (1100 IU/d) and Group 3 receives both placebos.

A full-service market research firm randomly selected telephone numbers from all households with listed numbers in the nine-county rural sample area. The firm continued calling until 1180 women were selected who met the inclusion and exclusion criteria and were willing to participate in a four year prospective study of calcium and vitamin D supplementation. The participants were enrolled into study between May 2000 and July 2001.

Participants have study visits every six months. Annually the following are performed: bone density scans, height and weight, brief medical history including medicine changes, fracture surveillance, and compliance with calcium and vitamin D. At baseline and end of study, spine x-rays and dietary recall were obtained.

ELIGIBILITY:
Inclusion Criteria: healthy women ages 55 and older who were at least four years postmenopausal living independently in a nine-county rural area of Nebraska

-

Exclusion Criteria:

1) chronic kidney disease, 2) Paget's metabolic bone disease, and 3) history of cancer except for superficial basal or squamous cell carcinoma of the skin and

-

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2000-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
fractures | 4 years

SECONDARY OUTCOMES:
changes in bone mass and density | 4 years
changes in serum dihydroxyvitamin D | one year and four years
changes in serum parathyroid hormone | one year and four years
cancer | four years
Falls | four years

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Lappe, Ph.D, Principal Investigator — Creighton University

REFERENCES:
- [Result] Lappe JM, Travers-Gustafson D, Davies KM, Recker RR, Heaney RP. Vitamin D and calcium supplementation reduces cancer risk: results of a randomized trial. Am J Clin Nutr. 2007 Jun;85(6):1586-91. doi: 10.1093/ajcn/85.6.1586. PMID 17556697
- [Derived] Zhou Y, Zhao LJ, Xu X, Ye A, Travers-Gustafson D, Zhou B, Wang HW, Zhang W, Lee Hamm L, Deng HW, Recker RR, Lappe JM. DNA methylation levels of CYP2R1 and CYP24A1 predict vitamin D response variation. J Steroid Biochem Mol Biol. 2014 Oct;144 Pt A:207-14. doi: 10.1016/j.jsbmb.2013.10.004. Epub 2013 Oct 12. PMID 24128439